CLINICAL TRIAL: NCT04554615
Title: Intensive Insulin Therapy as Therapeutic Strategy for Non-diabetic Hyperglycemia After Surgery in ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, MOHAMMED FAWZI ALI ABOSAMAK, Clinical professor of anesthesia and critical care, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Postoperative hyperglycemia
Record Dates: First submitted 2020-09-03; First posted 2020-09-18 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Hyperglycemia; Postoperative Complications; Insulin Resistance
MeSH Terms: conditions — Hyperglycemia; Postoperative Complications; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Insulin Therapy (Active Comparator): CIT was provided as a continuous infusion of 50 IU of Actrapid HM in 50 ml of 0.9% sodium chloride using a pump, Infusion was adjusted to achieve BG level in range of 180-200 mg/dl.
  Interventions: Drug: Insulin
- Intensive Insulin Therapy (Active Comparator): IIT was provided as an insulin infu-sion at rate of 1 mU/kg/min and was adjusted to achieve target BG level in range of 80-110 mg/dl.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — insulin infusion to control postoperative hyperglycemia
  Other Names: Blood sugar measurement

SUMMARY:
The current study hypothesizes that the use of Intravenous intensive insulin therapy (IV-IIT) may be beneficial than IV conventional insulin therapy (IV-CIT) for improving the outcome of non-diabetic surgical patients had postoperative (PO) stress hyperglycemia (PSH).

DETAILED DESCRIPTION:
All postoperative patients who will be admitted to surgical ICU and develop (PSH) will be eligible for evaluation for inclusion and exclusion criteria.

Prior to initiation of IV-IT (insulin therapy), blood samples will be obtained to estimate base-line Blood Glucose level (BG). BG will be estimated hourly during IV-IT to guard against development of hypoglycemic episodes. The assigned IV-IT will continue till reaching the target BG for each group and then will be stopped and patients will be shifted to subcutaneous (sc)-IT. During maintenance sc-IT, BG level will be estimated 6-hourly to assure maintenance of BG within the desired range, otherwise if hyperglycemia recurred or its induced complications as hyperglycemic ketoacidosis or hyperosmolar coma or infectious complications developed, IV-IT will be resumed and BG will be followed-up hourly. The same sequence of follow-up will be continued till stability of BG at the targeted level. IV-IT will be provided as following :

Conventional insulin therapy (CIT) will be provided as a continuous infusion of 50 IU of Actrapid HM in 50 ml of 0.9% sodium chloride using a pump. Infusion will be adjusted to achieve BG level in range of 180-200 mg/dl.

Intensive insulin therapy (IIT) will be provided as an insulin infusion at rate of 1 mU/kg/min and will be adjusted to achieve target BG level in range of 80-110 mg/dl.

ELIGIBILITY:
Inclusion Criteria:

* All postoperative patients who will be admitted to surgical ICU and developed Post Surgical Hyperglycemia will be eligible for evaluation for inclusion and exclusion criteria

Exclusion Criteria:

* All patients having diabetes mellitus, history of preoperative stress hyperglycemia, endocrinopathies, obesity defined as body mass index (BMI) >30 kg/m2, age younger than 18 years, renal impairment or maintenance on renal replacement therapy and liver diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2018-03-03 (Actual); Study Completion 2018-06-10 (Actual)

PRIMARY OUTCOMES:
The number of IV-Insulin Therapy sessions required till stabilization of the targeted Blood Glucose level. | 180 days
  insulin infusion will be given in shots to control the high blood sugar and the times of giving these shots will be counted

SECONDARY OUTCOMES:
Duration to control hyperglycemia | 180 days
  the duration till stabilization of the targeted BG level
28-day ICU morbidity | 180 days
  hyperglycemic hyperosmolar coma, diabetic ketoacidosis and infections will be documented.
28 - day ICU mortality | 180 days
  patients died within 28 days of ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abosamak, Principal Investigator — Tanta University
Locations (1):
- Security Forces Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
Once approved by clinical trial.gov data will be participated